CLINICAL TRIAL: NCT00172250
Title: The Study of Relationship of Plasma Concentrations of Folic Acid, Vitamin B and Homocysteine With Carotid Atherosclerosis and Endothelium-Dependent Vasodilatation of Geriatric and Young Patients in the Ambulatory Care Department of NTUH
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701046
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-08

CONDITIONS: Homocysteine; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Elevation of plasma homocysteine has been recognized as one of the risk factors of atherosclerotic disease. The objectives of this study are: (1) to investigate the level of plasma homocysteine and the prevalence of hypehomocysteinemia (2) to find out the role of homocysteine in coronary artery disease and the proper cut-off point of plasma homocysteine to evaluate the presence of coronary artery disease; (3) to understand the control condition of tranditional risk factors of cardiovascular disease, especially hypertension, dyslipidemia, and diabetes mellitus.

The study subjects were recruited from the ambulatory setting of cardiology in National Taiwan University Hospital.

ELIGIBILITY:
Inclusion Criteria:

Patient > 65 y/o or < 50y/o Scr<=1.5mg/dL

Exclusion Criteria:

* Scr> 1.5mg/dl pregnancy alcohoism

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Juey-Jen Hwang, MD, PhD, Principal Investigator — National Taiwan University Hospital